CLINICAL TRIAL: NCT01292785
Title: Effects of Sex Steroid Hormones on Human Brain Function, Structure and Connectivity: A Longitudinal Study Using 7 Tesla Ultrahigh-field Magnetic Resonance Imaging
Brief Title: Effects of Sex Steroid Hormones on Human Brain Function, Structure and Connectivity
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, A/Prof. PD Dr., Medical University of Vienna
Other Study IDs: P23021FWF
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Gender Identity Disorder
MeSH Terms: conditions — Gender Dysphoria | interventions — Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Transsexual: Female-to-Male and Male-to-Female Transsexuals receiving hormonal therapy
  Interventions: Drug: Hormones
- Healthy control subjects: receiving no hormonal therapy

INTERVENTIONS:
Drug: Hormones — FtM will receive
  * 1000mg testosterone undecanoate every 12 weeks (Nebido® 4ml i.m.), or alternatively 50mg testosterone transdermally (Testogel® 5g-bag per day) and
  * if menstruation still occurs, additionally either lynestrenol Orgametril® (2-3 tablets/day) or in some cases 0.075mg desogestrel (Cerazette®, 1 tablet/day).
  MtF will receive
  * 50mg cyproterone acetate daily (Androcur®)
  * estradiol 100µg transdermal therapeutic system (TTS) twice a week (Estradot®, Estramon®), especially if subjects age is > 40 years, or p.o. estradiol 2x2mg (Estrofem®) if subjects age is < 40 years; alternatively estradiol 0,75-1,5mg (1-2 hubs) transdermally (Estrogel-Gel®) and
  * 2,5mg alpha-5-reductase-inhibitor every 2nd day (Finasterid Actavis/ Arcana/ Aurobindo®) in case of extensive hair loss.
  Groups: Transsexual

SUMMARY:
This ultrahigh-field MRI study gives us the unique opportunity to measure changes in brain function and structure induced by long-term opposite-sex steroid hormone administration in transsexual subjects. Our aim is 1. to prove the influence of high-dose, long-term opposite-sex steroid hormone treatment on functional brain response in transsexuals. 2. to investigate the influence of hormone treatment on resting state functional connectivity and brain morphology. 3. to investigate differences between transsexuals and healthy control subjects in brain function and functional connectivity, brain morphology and structural connectivity. In this longitudinal study, transsexuals and healthy control subjects will undergo three 7 Tesla ultrahigh-field MRI scan sessions: 1. baseline (before hormone treatment), 2. after 4 weeks of treatment and 3. after 4 months of treatment.

ELIGIBILITY:
Inclusion criteria for transsexuals are:

* DSM-IV diagnosis of Gender Identity Disorder (DSM-IV: 302.85, 302.6; ICD-10: F64.9, F64.8) by a structured clinical interview (SCID)
* general health based on history, physical examination, ECG, laboratory screening, SCID
* willingness and competence to sign the informed consent form

Exclusion criteria for transsexuals are:

* severe neurological or internal diseases
* steroid hormone treatment within 2 months prior to inclusion (including birth control pill, phytohormones)
* treatment with psychotropic agents such as SSRIs
* any implant or stainless steel graft
* abnormal values in routine laboratory screening or general physical examination
* current substance abuse (determined using drug screening at the screening visit)
* pregnancy (determined at screening visit and first MRI scan)
* failure to comply with the study protocol or to follow the instructions of the investigating team.

Inclusion criteria for healthy controls are:

* general health based on history, physical examination, ECG, laboratory screening, SCID
* willingness and competence to sign the informed consent form

Exclusion criteria for healthy controls are:

* severe diseases
* any implant or stainless steel graft
* steroid hormone treatment within 2 months prior to inclusion (including birth control pill, phytohormones)
* abnormal values in routine laboratory screening or general physical examination
* current substance abuse (determined using drug screening at the screening visit)
* pregnancy (determined at screening visit and first MRI scan)
* failure to comply with the study protocol or to follow the instructions of the investigating team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Transsexuals urging sex reassignment in a clinical setting will be enrolled at the Unit for Gender Identity Disorder at the General Hospital in Vienna. 20 female-to-male (FtM) and 20 male-to-female (MtF) transsexuals will be asked to undergo this fMRI, MRI, DTI and resting-state functional connectivity study. Transsexual subjects are aged between 18 and 50 years old and free from hormone-treatment at baseline.
  40 healthy control subjects, matched for age, sex and sexual orientation to transsexual subjects will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
BOLD response to experimental fMRI paradigms | at baseline, 1 and 4 months after treatment start
  task-related BOLD (blood oxygen level dependent) responses are evaluated before, and 4 weeks, as well as 4 months of hormonal treatment in transsexual subjects and healthy control subjects

SECONDARY OUTCOMES:
Psychological Questionaires | at baseline, 1 and 4 months after treatment start
  Psychological questionaires measuring different aspects of emotion and cognitive processing are used to infer effects of hormonal therapy on these measures

CONTACTS AND LOCATIONS:
Overall Officials: Rupert R Lanzenberger, A/Prof. MD, Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.meduniwien.ac.at/neuroimaging/